CLINICAL TRIAL: NCT06311708
Title: Seroprevalence Study of Pre-existing Antibodies Against Adenovirus-associated Virus Vector (AAV9) in Patients With Plakophilin 2 (PKP2)-Associated Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
Brief Title: Non-interventional Study of Seroprevalence of Pre-existing Antibodies Against Adenovirus-associated Virus Vector (AAV9) and the Progression of Disease in Patients With Plakophilin 2 (PKP2)-Associated Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
Acronym: RIDGE
Status: Recruiting | Type: Observational
Sponsor: Tenaya Therapeutics (Industry)
Collaborators: University of California, San Francisco (Other); Brigham and Women's Hospital (Other); New York University (Other); University of Colorado, Denver (Other); Johns Hopkins University (Other); The Cleveland Clinic (Other); Mayo Clinic (Other); Medical University of South Carolina (Other); Hopital Louis Pradel (Other); Istituti Clinici Scientifici Maugeri SpA (Other); The Queen Elizabeth Hospital (Other); St George's University Hospitals NHS Foundation Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); Skane University Hospital (Other); Centro Cardiologico Monzino (Other); Hôpital Haut-Lévêque (Other); Nantes University Hospital (Other); Pitié-Salpêtrière Hospital (Other); Wuerzburg University Hospital (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: TN-401-0011
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: PKP2 Mutation Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC); Arrhythmogenic Cardiomyopathy (ACM); PKP2-associated ARVC; PKP2-ARVC; PKP2-ACM; Adeno Associated Virus (AAV); Adeno-Associated Virus Serotype 9 (AAV9); Gene Therapy; Gene Transfer; Genetic cardiomyopathy; Heart Failure
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be collected throughout the study 1 time each year to assess proteins and biomarkers associated with ARVC and to study existing antibodies to AAV9.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective and Prospective: Patients who meet the eligibility criteria are observed and data collected both prospectively and retrospectively.

SUMMARY:
This is a multicenter, non-interventional study to observe the natural progression of the disease and to study the prevalence of pre-existing antibodies to AAV9 used for gene therapy in a population of patients with PKP2 gene-associated ARVC. Participation from all patients is encouraged regardless of interest in or eligibility for gene therapy.

DETAILED DESCRIPTION:
Patients will receive standard of care treatments and assessments under the care of their healthcare provider. Biologic samples will be collected annually to measure cardiac and other related biomarkers. Clinical and observational data will be collected prospectively for up to 5 years from the date of enrollment, or until the patient withdraws consent/assent, undergoes heart transplantation, or dies.

If consent is provided, there may be a one-time sample collection to evaluate genetics for research purposes. Quality of Life (QoL) questionnaires will be used to assess a patient's wellbeing and quality of life. If not included as part of a patient's standard of care, diagnostic Holter (or equivalent) monitoring will be required annually. No investigational product will be administered. Participation from all patients is encouraged regardless of interest in or eligibility for gene therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-65 years, inclusive, at the time of consent
* Pathogenic or likely pathogenic PKP2 gene mutation
* Diagnosed with ARVC and meet 2010 Modified Task Force Criteria for ARVC as affected.
* Functioning ICD

Exclusion Criteria:

* Currently receiving systemic immunosuppressive therapy, cytotoxic chemotherapy, immunoglobulin therapy or monoclonal antibody therapy
* History of clinically significant liver disease, hepatitis B virus, hepatitis C virus, human immunodeficiency virus, or tuberculosis infection
* Previously dosed with any investigational or approved gene therapy product at any time
* Concurrent participation in another interventional clinical trial unless approved by the Sponsor. Participation in a noninterventional study may be allowed at the investigator's discretion.
* History of cardiac transplant.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are 14-65 years of age at the time of consent, and with confirmed mutations in PKP2 gene with a diagnosis of ARVC.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2030-03-29 (Estimated); Study Completion 2030-07-11 (Estimated)

PRIMARY OUTCOMES:
Investigate the seroprevalence of pre-existing antibodies to AAV9 in patients with PKP2-associated ARVC | 5 years

SECONDARY OUTCOMES:
To characterize the burden of illness in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years
To characterize arrhythmic risk in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years
To evaluate functional status and Quality of Life (QoL) in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years
To evaluate heart function as assessed by imaging in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years

OTHER OUTCOMES:
• To monitor biomarkers associated with disease progression and inflammation in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years
To evaluate genetics associated with PKP2-associated ARVC | 5 years
To evaluate the effect of other cardiac mutations or other genetic variants that might affect the penetrance and/or expressivity of PKP2 mutations in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years
To evaluate health care utilization in patients with pathogenic or likely pathogenic PKP2 mutations | 5 years

CONTACTS AND LOCATIONS:
Locations (21):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
- France (4):
  - Hopital Louis Pradel, Bron
  - Nantes University Hospital, Nantes
  - Pitié-Salpêtrière Hospital, Paris
  - Hôpital Haut-Lévêque, Pessac
- Germany (2):
  - University Hospital Muenster, Münster
  - Wuerzburg University Hospital, Würzburg
- Italy (2):
  - Centro Cardiologico Monzino, Milan
  - Istituti Clinici Scientifici Maugeri SpA, Pavia
- Skåne University Hospital, Malmo, Sweden
- United Kingdom (4):
  - The Queen Elizabeth Hospital, Glasgow
  - Barts & The London Health NHS Trust, London
  - St. George's University Hospitals NHS Foundation Trust, London
  - Royal Brompton & Harefield NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No